CLINICAL TRIAL: NCT01612299
Title: Effects of Zortress® + Tacrolimus vs. Standard Immunosuppression on Progression of Coronary Artery Calcifications and Bone Disease in de Novo Renal Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was withdrawn for this study by the sponsor.
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Hartmut Malluche, MD, Professor and Chief, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3048108907
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Immunosuppression (Active Comparator): Tacrolimus + Myfortic®/Cellcept + Corticosteroids
  Interventions: Drug: Zortress® /Everolimus
- Zortress® (Experimental): Tacrolimus + Zortress® + Corticosteroids
  Interventions: Drug: Zortress® /Everolimus

INTERVENTIONS:
Drug: Zortress® /Everolimus — Standard immunosuppression: THY 1-1.5 mg/kg/d qd for a total of 6 mg/kg •TAC trough targets 0-3 mo 8-12 ng/ml 4-6 mo 6-10 ng/ml >6 mo 5-8 ng/ml•Myfortic® or CEL 360mg or 500mg po BID, and receiving THY then Myfortic® or CEL 720 mg or 1000mg PO BID once THY induction completed• COR 500mg MET IV pre-op,125mg MET IV q24h x 2 doses (Post-Op Days 1 &2) 20mg Pred PO daily x 2 wks 15mg Pred PO daily x 2 wks 10mg Pred PO daily x 4 wks 5mg Pred PO daily x 4 wks 5 mg Pred PO every other day through mon 12.
  Experimental: TAC + Zortress® + COR In this arm patients will stop Myfortic®/CEL and start Zortress® at a dose of 1 mg PO BID with a target level of 3-8 ng/ml.At Zortress® level of at least 3 ng/ml TAC will be dosed to a target range as follows Randomization through mo 3 post-transplant 7-10 ng/ml 4-6 mo post transplant 5-8 ng/ml >6 mo post transplant 4-7 ng/ml.

SUMMARY:
Primary objectives: A. To evaluate the effect of Zortress® versus standard immunosuppression therapy on progression of CAC as evidenced by changes in Agatston scores from baseline and at 6, and 12 months in renal transplantation patients. B. To investigate progression of CAC in patients undergoing renal transplantation within the study period.

Secondary objectives:

1. To evaluate in renal transplantation the effect of Zortress® versus standard immunosuppression therapy on bone mass as evidenced by changes in quantitative computed tomography (QCT) and dual energy X-ray absorptiometry (DXA).
2. To evaluate in renal transplantation the effect of Zortress® versus standard immunosuppression therapy on activity of bone forming and resorbing cells as evidenced by changes in bone histology.
3. To evaluate in renal transplantation the effect of Zortress® versus standard immunosuppression therapy on biochemical parameters of bone turnover as evidenced by changes in serum Parathyroid Hormone (PTH), Bone-Specific Alkaline Phosphatase (BSAP), Tartrate-Resistant Acid Phosphatase (TRAP), Sclerostin, Receptor Activator of Nuclear factor Kappa B Ligand (RANKL), Osteoprotegerin (OPG), , serum CTX (C-terminal telopeptide of type 1 collagen), and urinary NTX (N-terminal cross link telopeptide).
4. To evaluate in renal transplantation the effect of Zortress® versus standard immunosuppression therapy on cardiovascular events, graft rejection and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* De novo renal transplant recipients (from deceased or living donors) between 18-70 years of age
* Willingness to participate in the study and comply with study requirements as evidenced by signed IRB-approved informed consent

Enrollment Exclusion Criteria:

* Previous solid organ transplant
* Known hypersensitivity to any of the study drugs, or their class, or to any of their excipients
* Recipients of an investigational drug within 30 days before transplant
* Any abnormal physical or laboratory findings of clinical significance which would interfere with conduct of the study
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, or unwilling to use medically approved means of contraception

Randomization Exclusion Criteria:

* Platelet count <75,000/mm
* White blood cell count of < 2,000/mm³
* Hypercholesterolemia (>400 mg/dL) or hypertriglyceridemia (>500 mg/dL) despite lipid-lowering therapy
* Presence of any clinically significant infection requiring IV antibiotics
* Positive serum HCG (women of childbearing potential)
* Spot urine protein to creatinine ratio (UPr/Cr ) ≥ 0.5
* Any biopsy-confirmed acute rejection since transplant
* Baseline CAC score < 100 at baseline reading

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
progression of Coronary Artery Calcification | 1 year
  The primary outcome of this study is the proportion of pts in the treatment group who experience a 1yr increase of ≥2.5 for the square-root transformed volume indicating CAC progression. Student's Fisher's Exact T-tests will be used to determine progression of CAC score between control & treatment groups. Secondary objectives 1-3 examine 1yr changes in several measurement outcome variables. Fisher's exact tests & confidence intervals for the difference in proportions will be used to compare the two groups in terms of cardiovascular events, graft rejection, & pt survival.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Malluche, MD, Principal Investigator — University of Kentucky; Roberto Gedaly, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States